CLINICAL TRIAL: NCT05272644
Title: Efficacy of Biofeedback-Assisted Pelvic Muscle Floor Training and Electrical Stimulation on Women With Different Pathophysiological Classifications of Stress Urinary Incontinence
Brief Title: Efficacy of Biofeedback-Assisted Pelvic Muscle Floor Training and Electrical Stimulation on Women With Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109184-F
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Stress Urinary Incontinence; Urethral Hypermobility; Intrinsic Sphincter Deficiency
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: A total of 128 women with stress urinary incontinence will be divided into two groups: urethral hypermobility and intrinsic sphincter deficiency; and they will be further randomized to 2 arms: surface electromyographic biofeedback arm, surface electromyographic biofeedback and electrical stimulation arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- urethral hypermobility-surface electromyographic biofeedback only (Active Comparator): Participant will be doing surface electromyographic biofeedback assisted pelvic floor muscle training for 2 months
  Interventions: Behavioral: surface electromyographic biofeedback assisted pelvic floor muscle training
- urethral hypermobility-surface electromyographic biofeedback and electrical stimulation (Experimental): Participant will be doing surface electromyographic biofeedback and electrical stimulation assisted pelvic floor muscle training for 2 months
  Interventions: Behavioral: surface electromyographic biofeedback and electrical stimulation
- intrinsic sphincter deficiency-surface electromyographic biofeedback only (Active Comparator): Participant will be doing surface electromyographic biofeedback assisted pelvic floor muscle training for 2 months
  Interventions: Behavioral: surface electromyographic biofeedback assisted pelvic floor muscle training
- intrinsic sphincter deficiency-surface electromyographic biofeedback and electrical stimulation (Experimental): Participant will be doing surface electromyographic biofeedback and electrical stimulation assisted pelvic floor muscle training for 2 months
  Interventions: Behavioral: surface electromyographic biofeedback and electrical stimulation

INTERVENTIONS:
Behavioral: surface electromyographic biofeedback assisted pelvic floor muscle training — participants will be doing surface electromyographic biofeedback assisted pelvic floor muscle training for 2 months
  Arms: intrinsic sphincter deficiency-surface electromyographic biofeedback only; urethral hypermobility-surface electromyographic biofeedback only
Behavioral: surface electromyographic biofeedback and electrical stimulation — participants will be doing surface electromyographic biofeedback and electrical stimulation assisted pelvic floor muscle training for 2 months
  Arms: intrinsic sphincter deficiency-surface electromyographic biofeedback and electrical stimulation; urethral hypermobility-surface electromyographic biofeedback and electrical stimulation

SUMMARY:
The pathophysiological mechanism of stress urinary incontinence divides stress urinary incontinence into urethral hypermobility and intrinsic sphincter deficiency. Pelvic floor muscle exercise as first line therapy has been found to be extremely helpful in patients with mild to moderate forms of incontinence. Biofeedback uses an instrument to record the biological signals ( electrical activity) during a voluntary pelvic floor muscle contraction and present this information back to the woman in auditory or visual form. Electrical stimulation can aid in detecting pelvic floor muscles, and also promote the contraction of the pelvic floor muscles and strengthen the muscles. This study assumes that urinary incontinence women with different pathophysiological classifications receiving a pelvic floor muscle training with surface electromyographic biofeedback and electrical stimulation show differences in the strength of pelvic muscle and degree of symptoms improvement.

DETAILED DESCRIPTION:
Participant will be assigned randomly to biofeedback-assisted pelvic floor muscle training (PFMT) group and biofeedback-assisted pelvic floor muscle training (PFMT) combined with electrical stimulation group. Each of the participant will receive the therapy for two months.The investigators expected that combination therapy will improve the compliance and severity of symptoms in women with stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. overactivity bladder for more than 3 months
2. more then 20 year old,less then 85 year old and acceptable to receive vaginal examination
3. need to match schedule with the investigator's clinic for 45 times,followed by individual therapy, each takes about 30 to 60 minutes, a total of 8 weeks of pelvic floor muscle exercises

Exclusion Criteria:

1. Suffering from systemic neuromuscular diseases, such as stroke, spinal cord injury, peripheral neuropathy, etc.
2. Kidney disease
3. Liver disease
4. Patients with cardiac rhythm devices.
5. Insufficient cognitive function, unable to cooperate with pelvic floor muscle exercises.
6. Women during pregnancy.
7. Maternity within six weeks after delivery

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
King's Health Questionnaire (KHQ) | Time Frame: through study completion, an average of 8 weeks
  KHQ has 3 parts consisting of 21 items. Part 1 contains general health perception and incontinence impact (one item each). Part 2 contains role limitations, physical limitations, social limitations (two items each), personal relationships, emotions (three items each) and sleep/energy (two items), severity measures (four items).Part 3 is considered as a single item and contains ten responses in relation to frequency, nocturia, urgency,urge, stress, intercourse incontinence, nocturnal enuresis,infections, pain, and difficulty in voiding. The 4 subscales scored between 1 (best) and 4 (worst) in part 1 and 2. The Symptom Severity scale is scored from 0 (best) to 3 (worst) in part 3 .
A five-item Self-Assessment of Treatment (SAT) | Time Frame: through study completion, an average of 8 weeks.
  to assess improvement and satisfaction with treatment, consists of 1 item. The scale scored between 1 (worst) and 5 (best ) .
Sandvik urinary incontinence severity test | Time Frame: through study completion, an average of 8 weeks
  The Sandvik test was developed by Sandvik et al to be used as a simple way to calculate severity of urinary incontinence in women. Answer the two questions below and your result will be displayed (Severity Index Score).
Symptom Indexes for Stress Incontinence | Time Frame: through study completion, an average of 8 weeks
  assigning a grade based on a clinical history of incontinence: grade 1-only on Severe coughing, sneezing, lifting heavy objects, lifting heavy objects, jumping; grade 2-on walking or running; grade 3-on walking, doing housework (eg washing dishes, sweeping the floor), changing posture (eg from standing to squatting or sitting...);grade 4-on Resting state, such as turning over in bed

SECONDARY OUTCOMES:
Introital and transvaginal ultrasound in the assessment of urogenital and pelvic floor dysfunction | Time Frame: through study completion, an average of 8 weeks
  the transducer is placed over the external urethral orifice with the transducer axis corresponding to the body axis Ultrasound assessment of the bladder and urethra starts in the midsagittal plane.
  From this position, the transducer can be moved to the left or to the right for additional assessment of the periurethral tissue. The distance between bladder neck and line through the lower edge of the pubic symphysis, and the posterior urethrovesical angle β (angle between urethral axis and bladder floor) are determined at rest and during contraction, coughing, and pressing. Changes in these parameters during contraction and pressing and in particular visual real-time ultrasound assessment serve to evaluate the reactivity of the pelvic floor muscles and the adequacy of the connective tissue supportive structures of the urogenital organs.
one-hour pad test | Time Frame: through study completion, an average of 8 weeks
  The test is carried out according to the recommendations of the International Continence Society and lasts for one hour and fifteen minutes. It consists in weighing the amount of urine retained in a sanitary napkin after the patient has completed a set of standard exercises, distributed over an hour.
change of electromyographic activity | Time Frame: through study completion, an average of 8 weeks
  Electromyographic activity of the pelvic floor muscles (PFMs) and the synergistic abdominal muscles (SAMs) during each session of PFMT(µV)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan